CLINICAL TRIAL: NCT03989661
Title: Is There a Place for Pre-operative Temporary Embolization of Uterine Fibroids
Acronym: EMBOFIB
Status: Completed | Type: Observational
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: EMBOFIB
Record Dates: First submitted 2019-06-14; First posted 2019-06-18 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2022-04

CONDITIONS: Uterine Fibroid
MeSH Terms: conditions — Leiomyoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Test group: This group corresponds to patients who had undergone preoperative embolization (with resorbable material) before myomectomy.
- Control group: This group corresponds to patients with myomectomy without embolization.

SUMMARY:
Uterine fibroids are the most common benign tumors of the female genital tract, with an estimated incidence of 25-80% during the reproductive period in the general population.

If the affected patients do not usually have any symptoms, uterine fibroids may also, depending on their location, be responsible for acute and chronic pelvic pain, bleeding and infertility.

Symptomatic uterine fibroids are now treated in the first line by surgery (hysterectomy, laparotomy myomectomy, laparoscopy or hysteroscopy). When conservative treatment is indicated and the fibroid is not hysteroscopically accessible, myomectomy can be performed by laparotomy or laparoscopy.

Excision of myomas often richly vascularized exposes the surgeon and the patient to a risk of bleeding per- and / or post-operative sometimes severe, resulting in an increase in operating times, an increased risk of postoperative complications and need transfusion.

The literature is rather poor on this subject but some factors favoring bleeding have been identified: the history of myomectomy, a uterine volume equivalent to more than 20 weeks of amenorrhea, the excision of more than 10 fibroids, or an incisional approach.

In order to reduce these intraoperative bleeds, numerous therapeutic strategies have been developed, using drug alternatives (GnRH agonists, Ullipristal) or interventional radiology (embolisation of the uterine arteries).

The improvement of interdisciplinary collaboration is now seeing the emergence of numerous therapeutic strategies combined.

The effectiveness of uterine artery embolization has been demonstrated for several years in the treatment of fibroids, alone or in combination with surgical myomectomy.

Some studies on preoperative embolization (maximum 24 hours before the intervention) have shown encouraging results with regard to the volume of bleeding, the need for per or post-operative transfusion or the need for surgical revision, or even decision to hystérectomie.

In 2011, Butori et al. propose the use of absorbable spongy particles (Curaspon type) for preoperative embolization. The use of these resorbable particles would reduce the risk of postoperative synechia. Some studies indicate that embolization of the uterine arteries using non-absorbable material would be responsible for ovarian failure by hypo-infusion. The use of absorbable material would avoid this adverse effect while preserving its effectiveness for the surgical procedure, but to date no study clearly demonstrates this.

This retrospective case-control study aims to compare the occurrence of per-and post-operative adverse effects between a test group consisting of patients who had undergone preoperative embolization (with resorbable material) before myomectomy (intervention group) and a control group with myomectomy without embolization (control group).

ELIGIBILITY:
Inclusion Criteria:

* Patients whose age is ≥ 18 years
* Patients who underwent a single myomectomy or laparotomy polymyomectomy in the gynecological surgery department of the Paris Saint-Joseph Hospital Group between January 2016 and June 2018, with or without preoperative embolization
* Francophone patients

Exclusion Criteria:

* - Patients under guardianship or curatorship
* Patient deprived of liberty
* Patient opposing the use of his data for this research

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent a single myomectomy or laparotomy polymyomectomy in the gynecological surgery department of the Paris Saint-Joseph Hospital Group between January 2016 and June 2018, with or without preoperative embolization
Sampling Method: Non-Probability Sample
Enrollment: 119 (Actual)
Dates: Start 2019-07-12 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Risk of intraoperative hemorrhage | Day 1
  This outcome measure pre- and postoperative hemoglobin levels for the 2 groups.

SECONDARY OUTCOMES:
Intraoperative transfusion rate | Day 1
  This outcome measure the number of patients who had Intraoperative transfusion.
Post-operative transfusion rate | Day 1
  This outcome measure the number of patients who had post-operative transfusion.

CONTACTS AND LOCATIONS:
Overall Officials: Eric SAUVANET, MD, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (1):
- Groupe Hospitalier Paris Saint-Joseph, Paris, France